CLINICAL TRIAL: NCT04772547
Title: VIGABatrin in Post-anoxic STATus Epilepticus - Phase IIa
Acronym: VIGAB-STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Yale University (Other); Thomas Jefferson University (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIGAB-STAT IIa; IRB202003076 (Other: UF IRB-01); OCR40379 (Other: UF OnCore); PRO00031111 (Other: UFIRST); 20IPA35380013 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Status Epilepticus, Electrographic; Coma
Keywords: post-anoxic status epilepticus, cardiac arrest, nonconvulsive status epilepticus, coma, vigabatrin
MeSH Terms: conditions — Status Epilepticus; Coma; Heart Arrest | interventions — Vigabatrin

STUDY DESIGN:
Intervention Model Description: pilot feasibility trial of pharmacokinetics of drug absorption
Masking Description: Participants are unconscious, thus, inherently blinded to the intervention. All the endpoints are objective and will be assessed by a blinded investigator to the timing of vigabatrin administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental): 4500 mg of vigabatrin administered enterally
  Interventions: Drug: Vigabatrin Only Product

INTERVENTIONS:
Drug: Vigabatrin Only Product — enteral medication administration, serial blood draws, and outcome assessment
  Other Names: sabril, vigabatrone

SUMMARY:
This is a pilot trial of a single loading dose of vigabatrin in post-anoxic status epilepticus.

DETAILED DESCRIPTION:
This pilot trial aims to demonstrate the feasibility of enteral administration of a single load of vigabatrin within targeted 48 hours of post-anoxic status epilepticus onset in unconscious survivors of cardiac arrest undergoing targeted temperature management. The load of VGB is in addition to the load of a commonly used intravenous second-line therapy given at the discretion of the treating neurologist. Serial blood tests will be obtained, including vigabatrin levels, taurine levels, neuron specific enolase, light chain neurofilament, and glial fibrillary acidic protein. In survivors that regain consciousness and survive to follow up, 6 months visual field perimetry will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* non-traumatic cardiac arrest (regardless of non-perfusing rhythm, etiology, or location of arrest) in whom the decision to treat unequivocal electrographic status epilepticus (as defined by the American Clinical Neurophysiology Society: having generalized spike/sharp-wave discharges ≥ 3Hz or any evolving pattern reaching > 4Hz, lasting ≥ 10 minutes, or comprising > 50% of any hour of recording) has been made
* requiring anesthetic infusion for any reason
* have reliable arterial access for frequent blood sampling
* established enteral access within 48h of post-anoxic status epilepticus onset.

Exclusion Criteria:

* prior history of generalized epilepsy
* history of gastrointestinal surgery within the last 21 days
* pregnancy
* status epilepticus onset preceding initiation of electroencephalography monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina B Maciel, MD, MSCR, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maciel CB, Teixeira FJP, Dickinson KJ, Spana JC, Merck LH, Rabinstein AA, Sergott R, Shan G, Miao G, Peloquin CA, Busl KM, Hirsch LJ. Early vigabatrin augmenting GABA-ergic pathways in post-anoxic status epilepticus (VIGAB-STAT) phase IIa clinical trial study protocol. Neurol Res Pract. 2022 Jan 24;4(1):4. doi: 10.1186/s42466-022-00168-x. PMID 35067230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment occurred from September 2021 until June 2023 at the University of Florida, Shands Hospital. All patients with cardiac arrest requiring continuous EEG (cEE) monitoring were screened for eligibility.
Pre-assignment Details: A total of 161 cardiac arrest patients requiring continuous EEG monitoring were screened for eligibility. Of the 8 patients deemed eligible, 75% (n=6) were enrolled.
Groups:
- Open Label: Vigabatrin administered enterally with serial blood draws and outcome assessment. Drug dose adjusted according to renal function.(CrCl>50 ml/min: 4500 mg; CrcL 30-50 ml/min: 2,250 mg; Crcl< 30 ml/min: 1,125 mg)
Period: Overall Study
Arm/Group | Open Label
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Vigabatrin administered enterally with serial blood draws and outcome assessment. Drug dose adjusted according to renal function.(CrCl>50 ml/min: 4500 mg; CrcL 30-50 ml/min: 2250 mg; Crcl< 30 ml/min: 1125 mg)
Arm/Group | Open Label
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.22 (13.11)
Creatinine Clearance (CrCl) [Count of Participants; unit: Participants]
  CrCl >50 ml/min | 2
  CrCl 30-50 ml/min | 2
  CrCl <30 ml/min | 2
Weight [Mean (Standard Deviation); unit: kg] | 88.03 (32.12)
Vigabatrin Dose Administered [Count of Participants; unit: Participants]
  4500 mg | 2
  2250 mg | 2
  1125 mg | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Pharmacologic Outcome - Absorption
Description: By analyzing serial vigabatrin levels including baseline, we characterized vigabatrin absorption; the target was to achieve a detectable vigabatrin level in the serum of ≥ 80% of enrolled subjects by 3 hours post-load.
Time Frame: 3h
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants
  Detectable drug level 3h post-administration | 6
  Undetectable drug level 3h post-administration | 0

2. Primary Outcome: Primary Feasibility Outcome - Enrollment and Drug Delivery
Description: We looked at the ability to deliver vigabatrin within 48 hours of PASE onset in ≥ 80% of enrolled subjects. Vigabatrin dose was adjusted according to renal functioning (CrCl>50 ml/min: 4500 mg, CrCl 30-50 ml/min: 2250 mg, CrCl<30 ml/min: 1125 mg)
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- Open Label: Vigabatrin administered enterally with serial blood draws and outcome assessment. Drug dose adjusted according to renal function.(CrCl>50 ml/min: 4500 mg; CrCl 30-50 ml/min: 2250 mg; CrCll< 30 ml/min: 1125 mg)
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants
  Vigabatrin administered within 48h of PASE onset | 6
  Vigabatrin not administered within 48h of PASE onset | 0

3. Primary Outcome: Primary Feasibility Outcome - Visual Screening (Goldmann Perimetry)
Description: We planned to obtain Goldmann perimetry testing in the subjects who could cooperate at the 6 months follow-up. Our goal was to have reliable visual field perimetry in ≥ 80% of survivors who regained consciousness following index hospitalization.
Time Frame: 6 months
Population: The 6 month follow-up could not be completed for any of the 6 enrolled subjects due to in-hospital mortality
Arm/Group | Open Label
Number analyzed (Participants) | 0

4. Primary Outcome: Primary Feasibility Outcome - Participants With Visual Screening for Taurine Levels
Description: We obtained serial taurine levels during ICU stay at time 0h, 72h and 168h following vigabatrin administration. Our goal was to achieve a 90% completion rate for taurine levels.
Time Frame: 0h, 72h and 168h following vigabatrin administration
Population: At the 72h timepoint following vigabatrin administration, data for only 5 of the six subjects was analyzed due to the death of one subject before the 72h timepoint. At 168h, data for only 2 of the six subjects was analyzed due to death of four subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants
  Taurine levels collected at 0h | 6
  Taurine levels collected at 72h: number analyzed (Participants) | 5
  Taurine levels collected at 72h | 4
  Taurine levels collected at 168h: number analyzed (Participants) | 2
  Taurine levels collected at 168h | 1

5. Secondary Outcome: Ultra-early Vigabatrin Administration
Description: We tracked the proportion of enrolled subjects who received a vigabatrin load within 12 and 24 hours of PASE onset to explore the possibility of ultra-early administration of vigabatrin in subsequent phases.
Time Frame: 0h to 48h after vigabatrin admnistration
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants
  within 12h of PASE onset | 1
  within 12-24h of PASE onset | 3
  within 24-48h of PASE onset | 2

6. Secondary Outcome: Secondary Pharmacologic Outcome: Elimination
Description: By analyzing serial VGB levels, we characterized drug elimination. We anticipated subjects with normal renal function would have undetectable vigabatrin levels by 72 hours, and those with creatinine clearance less than 30 mL/min would have detectable VGB levels at 72 hours. We anticipated undetectable vigabatrin levels in all subjects by 7 days regardless of their renal function.
Time Frame: 72h and 7 days following vigabatrin administration
Population: 72 hours after vigabatrin administration, vigabatrin concentration draws were done for only 4 of the 6 subjects, due to the death of 2 subjects. Both the subjects that died had CrCl<30 ml/min. All 4 of the subjects analyzed had CrCl>30 ml/min. Therefore, the results could not be stratified based on creatinine clearance level.
  7 days after vigabatrin administration, vigabatrin concentration draws were completed for only 2 of the six subjects, due to the death of the other 4 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 4
Participants
  Undetectable vigabatrin concentration at 72h | 2
  Detectable vigabatrin concentration at 72h | 2
  Undetectable vigabatrin concentration at 7 days: number analyzed (Participants) | 2
  Undetectable vigabatrin concentration at 7 days | 2
  Detectable vigabatrin concentration at 7 days: number analyzed (Participants) | 2
  Detectable vigabatrin concentration at 7 days | 0

7. Secondary Outcome: PASE Onset Detection
Description: We tracked the proportion of subjects in whom PASE was present upon connection to EEG (onset misses) to explore alternatives to allow prompt EEG monitoring following the return of spontaneous circulation (ROSC).
Time Frame: Determined at the time of connection to EEG monitoring
Population: The study did not enroll patients with PASE onset preceding the initiation of EEG monitoring. However, as a secondary exploratory outcome, we characterized the number of PASE-onset misses by determining the number of screen-failed patients, whose reason for screen failure was PASE onset preceding EEG monitoring initiation.
Measure: Count of Participants; unit: Participants
Groups:
- PASE Onset Misses: All cardiac arrest patients connected to cEEG monitoring screened for the trial.
Arm/Group | PASE Onset Misses
Number analyzed (Participants) | 161
Participants | 8

ADVERSE EVENTS:
Time Frame: As per clinical trial protocol, all subjects were monitored daily for adverse (AE) and serious adverse events (SAE) from the time of enrollment for the duration of their ICU stay. The PI monitored patient safety data within 24 hours of AE's or SAE's. The duration of ICU stay for the subjects was approximately 1 week. Screening for visual AE's was planned at the 6-month follow-up visit. Due to inpatient mortality, none of the enrolled subjects completed the 6-month follow-up.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
We could not characterize the exploratory safety outcome in our subjects. We aimed to detect rates of retinopathy on vision loss screening via Goldmann perimetry upon regain of consciousness, ICU discharge, and 6 months, in addition to long-term visual screening at 6 months via Visual Function Questionnaire 25 (VFQ-25). However, all six patients enrolled in the trial did not regain consciousness or survive through the follow-up period. So, the assessments could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT04772547/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04772547/ICF_001.pdf